CLINICAL TRIAL: NCT07019623
Title: Uro-catheter Vacuum-induced Uterine Tamponade (U-CaVIT) Versus Standard of Care for Prevention of Atonic Postpartum Hemorrhage After Cesarean Section in High-risk Women: a Monocentric Randomized-controlled Pilot Study.
Brief Title: U-CaVIT Versus Standard of Care for Prevention of Atonic Postpartum Hemorrhage After Cesarean Section in High-risk Women.
Acronym: UCaVIT Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Haslinger (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Christian Haslinger, Prof. Dr. med., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BASEC No. 2024-D0099
Record Dates: First submitted 2025-04-22; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Postpartum Hemorrhage (Primary); Hemorrhage; Postpartum Complication; Delivery ,Complications,Maternal; Pregnancy Complications; Cesarean Delivery; Balloon
Keywords: Postpartum Hemorrhage; Delivery complications; high risk patients; Pregnancy; Balloon Catheter; Tamponade; prophylactic; Vacuum-induced tamponade
MeSH Terms: conditions — Postpartum Hemorrhage; Hemorrhage; Pregnancy Complications | interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: This Investigator-initiated Trial (IIT) is a prospective, single-center, randomized-controlled study conducted in a prophylactic setting.
Who Masked: Outcomes Assessor
Masking Description: The analysis of the primary outcome will be performed using blinded treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- U-CaVIT (Experimental): Prophylactic treatment with Rüsch® Balloon Catheter Ch. 24
  Interventions: Device: Rüsch® Balloon Catheter Ch. 24; Other: Ultrasonography
- Control (No Intervention): Women in the control group will be treated according to the standard of care procedure.

INTERVENTIONS:
Device: Rüsch® Balloon Catheter Ch. 24 — After cesarean delivery, patients in the intervention group receive the following intervention: The Rüsch® Balloon Catheter Ch. 24 will be inserted directly into the uterus before uterotomy closure.
  After insertion of the catheter, the catheter balloon is filled with 60 - 80 ml of 0.9% saline solution and connected to the vacuum device whereby an intrauterine vacuum of -60 to a maximum of -70 kPa is applied once the uterotomy is closed. Once the catheter has been positioned, it is left in place for one hour as a prophylactic measure while a vacuum is applied.
  The device will be removed by draining the liquid in the balloon, after 1 hour of vacuum-induced tamponade. The final decision for removal of the catheter in this study is made by the senior physician responsible for the woman.
  Arms: U-CaVIT
Other: Ultrasonography — The position of the balloon catheter as well as the condition of the uterine cavity are assessed immediately postoperatively using ultrasonography.
  Arms: U-CaVIT

SUMMARY:
This pilot study aims to assess performance, safety and feasibility of U-CaVIT method (Uro-Catheter Vacuum Induced Tamponade), using the Rüsch® Brillant Silicone Balloon Catheter, an urological catheter, for the prevention of atonic PPH in high-risk women undergoing cesarean delivery.

The U-CaVIT method has been implemented at the Department of Obstetrics at university hospital of Zurich (USZ) due to temporary supply issues with the Bakri® Balloon Catheter. The Rüsch® Balloon Catheter is used in case of uterine atony when standard first-line uterotonic treatments have failed or in some cases as add-on therapy in non-atonic PPH. In the meantime, the use of U-CaVIT has become standard practice at the USZ for the treatment of atonic PPH, appearing to be user-friendly, clinically effective according to treating physicians, well tolerated by the treated women and cost-saving compared to the previously used Bakri® Balloon.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is the main reason for maternal peripartum mortality and morbidity. It poses a significant burden not just in developing countries but also in industrialized nations, where an upward trend in PPH-related problems is being observed.

According to the WHO, PPH is defined as blood loss of 500 mL or more within 24 hours after delivery, and it causes about 30% of maternal deaths worldwide. The internationally observed trend towards increased PPH-related morbidity and mortality is disturbing and demands new strategies in the prevention and treatment of PPH.

The underlying causes of PPH are uterine atony (Tonus), trauma (Trauma), placental disorders (Tissue), and coagulopathy/hemorrhagic diathesis (Thrombin) as well as disorder of the coagulation system which itself aggravates bleeding. Among these, uterine atony, which prevents mechanical hemostasis, is thought to be responsible for 60-80% of PPH cases and remains one of the most frequent causes of postpartum hysterectomy.

Therapy of uterine atony is based on the use of uterotonic drugs, nonsurgical approaches (e.g., uterine massage, intrauterine tamponade with an intrauterine balloon, vacuum device, or packing) as well as surgical therapies (e.g., repair of a deep laceration or tear in the uterus, cervix, or vagina; uterine artery ligation; curettage; uterine compression sutures; hysterectomy). A reasoned and sequential treatment approach is based on a multistage strategy that starts from less invasive interventions proceeding to more invasive methods. The strategic goal is to prevent severe PPH by implementing a minimally invasive, effective and low-cost method at an early stage of PPH or even before PPH might occur in high-risk patients, who inherently have an increased bleeding risk following a cesarean section. This would result in an enormous benefit to the patient in terms of morbidity and mortality as well as a consistent and judicious approach in the use of resources.

In an atonic uterus, vessels are not constricted and hemorrhage ensues, prompting first-line therapy. When medical management alone is deemed unsuccessful, balloon tamponade is currently the next treatment option added to control uterine atony. A balloon is placed within the uterus and inflated with sterile saline solution to put sustained pressure on the uterus from the inside. The Bakri® Balloon (Cook Medical) is currently the most commonly described intrauterine tamponade balloon device in the literature. By applying external pressure to the uterine walls for 12-24 hours, the uterus may then involute and regain normal tone. Although tamponade has been demonstrated to be effective in controlling hemorrhage in 87% (95% CI 84-90%) of atony-related cases, the mechanism of action of using outward pressure to control bleeding from uterine atony is counterintuitive if the ultimate goal is uterine contraction.

Recently, intrauterine vacuum devices have been introduced, offering a new mechanism for achieving hemorrhage control by applying low-level intrauterine vacuum to facilitate the physiological forces of uterine contractions, constrict myometrial blood vessels, and achieve hemostasis. Unlike the Bakri® Balloon, this device is not inflated but induces negative pressure in the uterine cavity, an approach called vacuum-induced tamponade. Purwosunu et al. conducted a proof-of-concept investigation involving 10 women. The rationale for creating negative pressure is that the vacuum extracts intrauterine blood and, by reducing uterine volume, promotes physiological uterine contraction, constricts the spiral arteries, and thus controls uterine atony.

In 2017, the Department of Obstetrics at USZ introduced another vacuum tamponade system, using a modified Bakri® balloon system (off-label use) to achieve intrauterine vacuum. According to the SOP at USZ, the balloon is filled with sterile fluid (60-80 mL) and connected with a vacuum-device applying a low-level intrauterine vacuum (-60 to a maximum of -70 kPa).

All women with primary PPH at the USZ, who were treated with vacuum-induced tamponade (i.e., with the modified Bakri® Balloon System) between March 2017 and June 2020, were analyzed. It was concluded that the vacuum-induced tamponade is an easy-to-use technique, and second, that vacuum-induced tamponade is associated with the highest success rate (defined as no need for additional interventional treatment such as surgical intervention or embolization of the pelvic arteries) in women with uterine atony.

Due to temporary worldwide supply difficulties of the Bakri® Balloon, the Rüsch® Balloon Catheter was introduced at USZ in June 2023 (also off-label use). As it is an urological catheter, this new approach was called U-CaVIT (Uro-Catheter Vacuum Induced Tamponade). It quickly gained favor among treating physicians due to its ease of use and apparent excellent performance. The use of the Rüsch® Balloon Catheter instead of the >20 times more expensive Bakri® Balloon, has become standard practice at the Department of Obstetrics for the treatment of atonic PPH: When indicated (i.e. when the standard uterotonic PPH treatment consisting of the administration of oxytocin or carbetocin followed by prostaglandins has failed, or when bleeding continues despite removal of the placenta or retained placental tissue), the Rüsch® Balloon Catheter is used according to the USZ internal SOP "Vakuuminduzierte Tamponade".

Given the substantial burden of PPH and its high mortality rates, especially in low-income countries, the development of low-cost yet highly effective methods such as U-CaVIT with the Rüsch® Balloon Catheter is crucial for improving maternal outcomes globally, extending beyond developed nations. To address this need, the investigators conduct this clinical trial to systematically evaluate the U-CaVIT approach (using the Rüsch® Balloon Catheter) as a prophylactic measure in high-risk post-cesarean section patients. Furthermore, this pilot clinical investigation will provide reliable data and pave the way for the competitive funding of a large-scale, national, multi-center pivotal study to evaluate the effect of this method in women at risk of PPH. The impact might be significant both in terms of patient outcomes and the reduction of PPH-related costs during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Maternal age ≥18 years
* Gestational age ≥34+0 weeks of pregnancy at day of delivery
* Vital pregnancy
* Delivery mode: planned cesarean delivery
* High-risk patient for PPH specified by the presence of at least one of the following characteristics: Previous PPH, obesity (BMI ≥30 kg/m2), high parity (patient who has had ≥4 previous births (live or stillborn) at ≥20 weeks of gestation), very advanced maternal age ≥45 years, multiple gestation, polyhydramnios (defined as amniotic fluid index > 25 cm or deepest amniotic fluid pocket > 8 cm) at admission to delivery, suspected fetal macrosomia (estimated fetal weight ≥ 4500g)

Exclusion Criteria:

* Insufficient language skills in German or English to understand and sign informed consent
* Participation in another interventional study
* Emergency cesarean section (incl. patients undergoing cesarean after failed vaginal delivery)
* Women with regular and painful contractions and women who do not have time for sufficient consideration
* Clinical situations in which vacuum-induced uterine tamponade is unlikely to be effective or is contraindicated: Uterine or vaginal anomalies (genital tract congenital anomalies), cesarean section due to placenta previa or suspected placenta accreta spectrum, suspected uterine rupture, injuries of the cervix or vagina, submucous or intramural uterine fibroids which are buldging into the uterine cavity, deep endometriosis
* Planned atony-prophylaxis with oxytocin due to contraindication for carbetocin
* Previous MMC-repair (myelomeningocele-repair)
* Clinical diagnosis of chorioamnionitis, sepsis
* Allergy to any component of the device
* Known and proven diagnosis of bleeding disorder or thrombophilia
* Known thrombocytopenia during second half of pregnancy with thrombocytes < 100 G/L
* Known anemia during second half of pregnancy with Hb<80 g/L

The following exclusion criteria will only be checked during the intra-operative assessment before randomization takes place:

* Cervix deemed too stiff and/or stenotic for U-CaVIT application, judged by the surgeon during the intra-operative assessment.
* Unexpected intraoperative findings incompatible with application of U-CaVIT (see above described clinical situations in exclusion criteria, in which vacuum-induced uterine tamponade is unlikely to be effective or is contraindicated).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in hemoglobin | From baseline (shortly before cesarean delivery) and 48 hours (range 36 to 60 hours) after cesarean delivery
  The primary outcome is to evaluate the postpartum change in hemoglobin (g/L) after cesarean delivery, comparing patients in the intervention group (treated with standard of care (SOC) plus U-CaVIT) to patients in the control group (treated with SOC).

SECONDARY OUTCOMES:
Postpartum hemoglobin (g/L) | Baseline (shortly before cesarean delivery) until hospital discharge (Follow-up 2), estimated 3 - 5 days after delivery
  Change of postpartum hemoglobin (g/L): Difference between prepartum and postpartum levels at hospital discharge
Blood loss | 24 hours after delivery
  Blood loss (ml): Estimated blood loss within 24 hours and during secondary PPH (if applicable).
Further PPH treatment/intervention. | Hospital discharge (Follow-up 2), estimated 3 - 5 days after delivery
  Need for further PPH treatment/intervention
Surgical revision | 24 hours after delivery
  Second operation within 24 hours
Uterotonic medication, of blood, blood products or coagulation factors. | 24 hours after delivery
  Administration of additional uterotonic medication, of blood, blood products or coagulation factors.
Postoperative coagulum | Hospital discharge (Follow-up 2), estimated 3 - 5 days after delivery
  Presence and size of postoperative coagulum
Secondary PPH | Randomization and hospital discharge (Follow-up 2), estimated 3 - 5 days after delivery
  Rate of secondary PPH
Bishop score (cervix score) | Baseline
  Evaluation of preoperative Bishop score and association of preoperative Bishop score with intraoperative assessment.
  The Bishop score evaluates the dilation, effacement, position, consistency, and the fetal head's station in the pelvis. Each parameter is assigned points, with a total score ranging from 0 to 13. Cervical dilation, effacement, and station are scored from 0 to 3 points, whereas cervical position and consistency are scored from 0 to 2 points.

OTHER OUTCOMES:
Other outcomes: usability of U-CaVIT | Hospital discharge (Follow-up 2), estimated 3 - 5 days after delivery
  The usability of U-CaVIT will be assessed by the investigators. From 2 days post-procedure until hospital discharge, a patient survey will be conducted to assess a woman's sensations of safety, anxiety, distress, and insecurity, as well as to evaluate personal peripartum satisfaction and experiences with U-CaVIT treatment (if applicable), including measures of discomfort, pain, and other related factors.
Safety Outcome | Randomization and hospital discharge (Follow-up 2), estimated 3 - 5 days after delivery
  Incidence of device-related serious adverse events, critical non-serious adverse events and device deficiencies.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Prof. Dr. med. Christian Haslinger, MD, Principal Investigator — University Hospital Zürich, Switzerland
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The data sharing plan aims to ensure computational reproducibility of all published research findings obtained from data collected in this trial. Each publication will be accompanied by a dedicated compendium containing deidentified individual patient data necessary to independently reproduce the analyses presented in the corresponding publication. Such a compendium also contains information about the computer code that was used to generate figures, tables, and other statistical output. Distribution will be via a data repository following FAIR principles (such as zenodo.org).
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: At the time of publication
Access Criteria: Access will be provided without limitations. Data will be provided to allow independent computational reproducibility of already published results.

REFERENCES:
- [Background] Goffman D, Rood KM, Bianco A, Biggio JR, Dietz P, Drake K, Heilman E, Hopkins M, De Four Jones M, Katz T, Martin C, Prasad M, Smid MC, Wine KD, Ryan R, Yong C, Carney PI, Simhan HN. Real-World Utilization of an Intrauterine, Vacuum-Induced, Hemorrhage-Control Device. Obstet Gynecol. 2023 Nov 1;142(5):1006-1016. doi: 10.1097/AOG.0000000000005366. Epub 2023 Sep 13. PMID 37713322
- [Background] D'Alton ME, Rood KM, Smid MC, Simhan HN, Skupski DW, Subramaniam A, Gibson KS, Rosen T, Clark SM, Dudley D, Iqbal SN, Paglia MJ, Duzyj CM, Chien EK, Gibbins KJ, Wine KD, Bentum NAA, Kominiarek MA, Tuuli MG, Goffman D. Intrauterine Vacuum-Induced Hemorrhage-Control Device for Rapid Treatment of Postpartum Hemorrhage. Obstet Gynecol. 2020 Nov;136(5):882-891. doi: 10.1097/AOG.0000000000004138. PMID 32909970
- [Background] Purwosunu Y, Sarkoen W, Arulkumaran S, Segnitz J. Control of Postpartum Hemorrhage Using Vacuum-Induced Uterine Tamponade. Obstet Gynecol. 2016 Jul;128(1):33-36. doi: 10.1097/AOG.0000000000001473. PMID 27275795
- [Background] Haslinger C, Weber K, Zimmermann R. Vacuum-Induced Tamponade for Treatment of Postpartum Hemorrhage. Obstet Gynecol. 2021 Sep 1;138(3):361-365. doi: 10.1097/AOG.0000000000004510. PMID 34352848
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301